CLINICAL TRIAL: NCT02363296
Title: Influence on Plasticity of Brain Temperature
Brief Title: Main Study: Influence on Plasticity of Brain Temperature Sub-Study: Phase Triggered Paired Associative Stimulation (PAS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 150066; 15-M-0066
Record Dates: First submitted 2015-02-13; First posted 2015-02-16 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09-30

CONDITIONS: Healthy Volunteers
Keywords: Paired Associative Stimulation; Brain Cooling (Main Study); Brain Cooling Helmet (Main Study); Repetitive TMS (rTMS); EEG phase-triggered TMS

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- EEG phase-triggered PAS (Experimental): TMS triggered to a specific phase of the EEG mu rhythm
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — Paired associative stimulation and single pulse TMS

SUMMARY:
Sub-Study: Phase Triggered Paired Associative Stimulation (PAS) (completed - analysis only)

Background:

-Previous research has shown that the brain s activity changes with changes in brain waves. We can study brain activity with a procedure called transcranial magnetic stimulation (TMS), a form of non-invasive brain stimulation. EEG allows for measuring ongoing brain waves. The goal of this study is to optimize TMS delivery by utilizing EEG-triggered TMS.

Objectives:

-To see if changes in brain waves change the brain and body s response to TMS.

Eligibility:

-Healthy, right-handed adults age 18-35.

Design:

* Participants will be screened under another protocol with medical history and physical exam. They may take a pregnancy test. They will have a magnetic resonance imaging (MRI) scan of the brain. For MRI, participants lie on a table that slides in and out of a metal tube that takes pictures. with:
* Participants will have up to 4 outpatient visits lasting 2-3 hours each (4 outpatient visits). The following procedures may occur at a visit:
* Magnetic resonance imaging (MRI): Participants lie on a table that slides into a machine that takes pictures of the brain.
* Electroencephalography (EEG): Small electrodes on the scalp record brain waves.
* Electromyography (EMG): Small sticky electrodes on the skin measure muscle activity.
* Transcranial magnetic stimulation (TMS): A wire coil is held to the scalp. A brief electrical current passes through the coil and affects brain activity.

Main Study: Influence on Plasticity of Brain Temperature (completed - analysis only)

Background:

- Brain activity changes with changes in body temperature. Brain activity can be studied with a procedure called transcranial magnetic stimulation (TMS). Researchers want to cool the brain through the scalp using a cooling cap. They want to see if cooling changes the brain and body s response to TMS.

Objectives:

- To look at the effects of cooling on the brain.

Eligibility:

- Right-handed adults age 18-50 who can abstain from caffeine and tobacco.

Design:

* Participants will be screened with medical history and physical exam. They will be asked about alcohol use, smoking, and substance abuse. They may take a pregnancy test. They may have a magnetic resonance imaging (MRI) scan of the brain. For MRI, participants lie on a table that slides in and out of a metal tube that takes pictures.
* Participants will have 3 outpatient visits. The following procedures will occur at each visit.
* Participants will wear a cooling cap for up to 45 minutes. Cool water will flow through the cap. It will feel like an ice pack in a towel. Their core temperature will be monitored. Their temperature will also be measured under their tongue and on scalp, stomach, forearm, and calf.
* Participants will have TMS before and after wearing the cap. A brief electrical current will pass through a wire coil held on their scalp. Electrodes that detect muscle movement will be placed on their hand. They will also have repetitive TMS, which uses repeated magnetic pulses. Their wrist will also receive a shock.

DETAILED DESCRIPTION:
1. Objective

   The dysregulation of synaptic transmission in certain brain areas may be responsible for some neurological disorders. It was demonstrated that synaptic transmission may be modulated through repetitive transcranial magnetic stimulation (rTMS), and this may be a component of the therapeutic effects of rTMS. However, rTMS utility is limited due to an inability to focus the stimulation and variability in intervention response. Cooling was shown to reduce the neuronal activity in targeted brain areas. The goal of this protocol is

   to examine the ability of cooling to affect rTMS.

   Sub-study: Phase-triggered paired associative stimulation (PAS)

   Similarly, response to transcranial magnetic stimulation (TMS) is variable. However, it has been demonstrated that EEG contains information impacting measurable TMS outcomes. The goal of this study is to optimize TMS delivery by utilizing EEG phase-triggered TMS.
2. Study population

   We intend to study 18 adult healthy volunteers on an outpatient basis. The accrual ceiling requested is 23 subjects to allow for dropouts and screening failures. This portion of the study has been completed and recruitment will not continue for the cooling-related

   portion of the study.

   Sub-study: Phase-triggered paired associative stimulation (PAS)

   We intend to perform a sub-study to develop a new method of plasticity induction- phase-triggered paired associative stimulation (PAS). This sub-study requires an additional intended study population of 24 subjects completing the 3 study arms who may be a sub-set of the initially requested 18 subjects from the main study. The additional accrual ceiling is 40 subjects to allow for dropouts and screening failures (24 participants complete sub-study/40 participants enrolled in sub-study). The total ceiling for the entire protocol is 63.
3. Design

   Analysis of the data collected during the main study demonstrates the control condition of rPAS/sham cooling did not result in increased motor evoked potentials (MEPs) as expected. This null effect of the control condition made it difficult to ascertain any effects due to the cooling condition. Therefore, we propose a new substudy investigating a better form of plasticity induction using EEG phase-triggered TMS.

   For the completed, cooling-related portion of the study, we propose using rapid-rate paired associative stimulation (rPAS), modulated by applying cooling to the scalp, to examine the effect of cooling on rTMS. Our hypothesis is that cooling the brain will prevent the potentiation normally induced by rPAS. We will reduce brain temperature by up to 1.5 degrees C by applying a cooling helmet to the scalp and then test the effect on potentiation by applying rPAS. One of our stopping criterion will be reduction in measured temperature reduction by 2 degrees C

   This study consists of one experiment with18 subjects and accrual has been completed. The experiment is divided into three session visits, each to be carried out at least 1 day apart.

   The control potentiation in response to rPAS without cooling will be measured during session visit 1 by using the TMS-evoked motor evoked potential (MEP). In session visit 2, after applying a commercially available liquid cooling helmet for 45 minutes to reduce the temperature of the underlying cerebral cortex by up to 1.5oC, we will then assess the response to rPAS. In session visit 3, the MEP will be measured after applying the cooling helmet but with the rPAS procedure substituted with a sham rPAS. Session visit 3 is necessary to determine if there are any changes to the MEP in response to cooling alone. Thus, in the three session visits, we will evaluate cooling alone, rPAS alone, and the two together.

   Sub-study: Phase-triggered paired associative stimulation (PAS)

   The proposed sub-study is to test a methodology to decrease the variability in response to and improve reliability of TMS, by utilizing EEG phase-triggered PAS. The new method will utilize EEG phase-triggered paired associative stimulation. Similarly to the rPAS used in the main study, EEG phase-triggered PAS also uses paired median nerve stimulation with TMS to motor cortex. However, the stimuli are triggered when the EEG recorded from the motor cortex (M1; EEGM1) is at a pre-specified phase of the alpha-band (8-12 Hz) oscillation.

   The sub-study to develop the optimal parameters of phase-triggered PAS will consist of upto 4 visits and 3 arms. The first visit is a screening and piloting visit, the subsequent visits are different arms of the study. Two active arms will trigger the paired median nerve and motor cortex TMS according to the phase of the ongoing EEG. One arm will trigger the stimuli at the trough of the ongoing EEG (phase -90 if the EEG is modeled as a sine wave). Another arm will trigger the stimuli at the peak of the ongoing EEG (phase +90). A control arm will trigger the paired stimuli at a random delay from the through of the ongoing EEG. This control arm serves to deliver paired stimuli at a rate matched to the ongoing EEG, but stimulates at a random phase of each alpha oscillation cycle. These arms will be pseudo-randomized.

   Our hypothesis is that stimulating at the through of the ongoing EEG will result in increased plastic changes to the brain as measured through our TMS outcome measures of single pulse MEPs, as compared to the control condition of random phase stimulation and stimulation at the peak of the ongoing EEG. We also hypothesize that stimulating at the peak of the ongoing EEG will result in a decrease in TMS outcome measures as compared to the control arm and stimulation at the trough of the ongoing EEG. This will be a within-subject design of 3 visits for each of the 40 sub-study subjects.
4. Outcome measures

The primary outcome measure will be the amplitude of MEPs induced by single TMS pulses.

Sub-study: Phase-triggered paired associative stimulation (PAS)

The primary outcome will be pre-post changes in MEP induced by phase-triggered TMS. Pre post changes in resting-state EEG (rs-EEG) will also be analysed. Associations between these outcomes and demographics will be included in the analyses.

ELIGIBILITY:
* INCLUSION CRITERIA:

Main Study:

To be eligible for this research study participants must:

* Be between 18 and 50 years of age.
* Be right-handed.
* Able to abstain from food or drinks containing caffeine 24 hours before the last 3 session visits. The screening visit does not require the ability to abstain from food or drinks containing caffeine.
* Able to abstain from tobacco on the day of the last three session visits. The screening visit doesn t require the ability to abstain from tobacco.

Sub-study: Phase-triggered paired associative stimulation (PAS)

* Males and females between 18 and 35 years of age.
* Subjects must be able to give written informed consent prior to participation in this study.

EXCLUSION CRITERIA:

Main Study:

Participants will be excluded from this research study if they:

* Are taking medications of the following classes: antidepressants, anxiolytics, anticonvulsants, antipsychotics, antiparkinson, hypnotics, stimulants, and antihistamines.
* Have a heart rate that exceeds 100 bpm (resting tachycardia).
* Have a history of psychiatric condition(s).
* Have a neurologic disorder such as a history of brain tumor, stroke, central nervous system infection, epilepsy, cerebrovascular disease, dementia, head trauma, or increased intracranial pressure.
* Have surgically or traumatically implanted metallic foreign bodies such as, pacemakers, medication pumps, implanted hearing aids, defibrillators, metal plates in the skull or metal implants in the skull or eyes (other than dental fillings), intracardiac lines, or any other condition/device that might be physically hazardous during TMS or magnetic resonance imaging (MRI), or might distort the images.
* Are unable to lie flat on back for up to 1 hour.
* Have claustrophobia or a feeling of discomfort from being in small, enclosed spaces of enough severity to prevent MRI scanning.
* Are pregnant or have a positive pregnancy test before the research procedure due to the risks associated with MRI scans and TMS.
* Have abnormal findings in clinical MRI that we will do during the screening visit.
* Have any abnormal or focal finding on the neurological exam.
* Have a known hearing loss.
* Have an alcohol or substance abuse problem, as determined by the Alcohol, Smoking and Substance Abuse Screening Test (ASSIST).
* Have sensitivity to coldness. (main experiment only, not an exclusion for the sub-study which does not utilize cooling)
* NIMH employees and staff and their immediate family members will be excluded from the study per NIMH policy.

Sub-study: Phase-triggered paired associative stimulation (PAS)

* Individuals taking medication that, in the opinion of the investigator, significantly lowers seizure threshold.
* Have a history of psychiatric condition(s).
* Have a neurologic disorder such as a history of brain tumor, stroke, central nervous system infection, epilepsy, cerebrovascular disease, dementia, head trauma, or increased intracranial pressure.
* Have abnormal findings in MRI that will be conducted during screening or prior to TMS under the current protocol
* Are pregnant or have a positive pregnancy test before the beginning of the study due to the risks associated with TMS.
* Subjects who have hearing loss that has been clinically evaluated and diagnosed.
* Any implant, prosthesis or other permanent alteration of the body that, in the opinion of the investigator, would be unsafe with TMS or that would produce an artifact that would compromise the integrity of data.
* Positive test for HIV.
* Have an alcohol or substance abuse problem.
* NIMH employees and staff and their immediate family members will be excluded from the study per NIMH policy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Motor evoked potential amplitude | immediate
  amplitude of motor evoked potentials recorded immediately after paired associative stimulation TMS.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zarate, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
An official plan has not been made as yet.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-M-0066.html